CLINICAL TRIAL: NCT07093567
Title: Opiophobia in Adults With Advanced Cancer
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0177; NCI-2025-05283 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the barriers and fears related to use of opioids among a population of adult outpatients with advanced cancer who continue to experience pain after receiving a prescription for opioid analgesia and hypothesized associations among opiophobia, anxiety, depression, pain intensity, pain interference, and opioid medication adherence.

DETAILED DESCRIPTION:
Primary Objective:

To explore the barriers and fears related to use of opioids among a population of adult outpatients with advanced cancer who continue to experience pain after receiving a prescription for opioid analgesia.

Secondary Objective:

To examine associations among opiophobia, anxiety, depression, pain intensity, pain interference, and opioid medication adherence among adults with advanced cancer who report undermanaged pain during the first week after receiving a prescription for an opioid analgesic.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with advanced cancer (defined as cancer that is unlikely to be cured and is locally advanced or distantly metastasized
2. Pain is the documented reason for the Supportive Care consultation
3. Have a prescription for an opioid analgesic
4. Able to read, speak, and consent in English.

Exclusion Criteria:

1. Age less than 18 years
2. Do not have a prescription for an opioid analgesic
3. Individuals for whom there is documentation of inability to provide consent in the medical record
4. Women who are pregnant
5. Patients with a substance use disorder (including alcohol use disorder and excluding tobacco use disorder) documented in the electronic health record under History of Present Illness or in the Medical History.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Barriers Questionnaire (BQ-13) | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Hacker, PHD, RN, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org